CLINICAL TRIAL: NCT03868163
Title: Real World Evidence of the Effectiveness and Clinical Practice Use of Glecaprevir Plus Pibrentasvir in Patients With Chronic Hepatitis C Genotypes 1 to 6 in Russian Federation
Brief Title: Real World Evidence of the Effectiveness and Clinical Practice Use of Glecaprevir Plus Pibrentasvir in Patients With Chronic Hepatitis C in the Russian Federation
Acronym: EVEREST
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-454
Record Dates: First submitted 2019-03-07; First posted 2019-03-08 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis C (CHC)
Keywords: Chronic Hepatitis C; Hepatitis C; Hepatitis; glecaprevir; pibrentasvir; real world setting; Observational Study
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Glecaprevir plus Pibrentasvir: Participants in this observational study will receive treatment with glecaprevir and pibrentasvir for up to 16 weeks for treatment of chronic hepatis C (CHC) genotypes 1, 2, 3, 4, 5, or 6.
  The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice, international guidelines and/or label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
This study seeks to assess the effectiveness of Glecaprevir plus Pibrentasvir in participants with chronic hepatitis C in a real-life setting across clinical practice populations in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or - pegIFN (or IFN), and/or Ribavirin (RBV) and/or sofosbuvir (PRS) experienced with confirmed CHC, genotypes 1, 2, 3, 4, 5, or 6, with or without compensated cirrhosis, receiving combination therapy with the all oral GLE/PIB regimen according to standard of care, international guidelines and in line with the current local label.
* May be enrolled up to 4 weeks after treatment initiation.
* Patients must voluntarily sign and date Informed Consent Form prior to inclusion into the study,
* Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CHC in a real world clinical practice setting.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12) | Up to approximately 28 weeks
  SVR12 defined as the hepatitis C virus (HCV) ribonucleic acid (RNA) level less than the lower limit of quantification/detection (<LLOQ/D) 12 weeks after the last dose of Glecaprevir plus Pibrentasvir (GLE/PIB).with a sensitive polymerase chain reaction [PCR] test with an LLoQ/D of <50 IU/mL or as described in a validated assay.

SECONDARY OUTCOMES:
Percentage of Participants Achieving SVR12 by Mono HCV or co-infected HCV/HIV Status | Up to approximately 28 weeks
  SVR12 defined as the HCV RNA level <LLOQ/D 12 weeks after the last dose of GLE/PIB.with a sensitive PCR test with an LLoQ/D of <50 IU/mL or as described in a validated assay.
Percentage of Participants Achieving SVR12 by CHC Genotype | Up to approximately 28 weeks
  SVR12 defined as the HCV RNA level <LLOQ/D 12 weeks after the last dose of GLE/PIB.with a sensitive PCR test with an LLoQ/D of <50 IU/mL or as described in a validated assay.
Percentage of Participants Achieving SVR12 by Cirrhosis Status | Up to approximately 28 weeks
  SVR12 defined as the HCV RNA level <LLOQ/D 12 weeks after the last dose of GLE/PIB with a sensitive PCR test with an LLoQ/D of <50 IU/mL or as described in a validated assay
Percentage of Participants Achieving SVR12 by Previous Treatment Experience | Up to approximately 28 weeks
  SVR12 defined as the HCV RNA level <LLOQ/D 12 weeks after the last dose of GLE/PIB with a sensitive PCR test with an LLoQ/D of <50 IU/mL or as described in a validated assay.
Percentage of Participants Achieving SVR12 by Patients Who Use Drugs | Up to approximately 28 weeks
  SVR12 defined as the HCV RNA level <LLOQ/D 12 weeks after the last dose of GLE/PIB with a sensitive PCR test with an LLoQ/D of <50 IU/mL or as described in a validated assay.
Percentage of Elderly Participants Achieving SVR12 | Up to approximately 28 weeks
  SVR12 defined as the HCV RNA level <LLOQ/D 12 weeks after the last dose of GLE/PIB with a sensitive PCR test with an LLoQ/D of <50 IU/mL or as described in a validated assay.
Percentage of Patients with Commodities | Up to approximately 16 weeks
  Percentage of Patients with Commodities from the decision to initiate treatment.
Percentage of Participants Taking Concomitant Medications | Up to approximately 28 weeks
  The percentage of participants taking concomitant medications from the decision to initiate treatment through up to 12 weeks after the last dose of GLE/PBR
Percentage of GLE/PIB Dose Taken | Up to approximately 16 weeks
  Percentage of GLE/PIB dose taken by patient report in relation to the prescribed target dose (that is, the number of pills taken out of the number that should have been taken).
Number of Health Care Resource Utilization (HCRU) | Up to approximately 28 weeks
  Health Care Resource Utilization (HCRU) for a patient will be the total number of visits/touchpoints (face to face or phone call) with a Health Care Provider (HCP) or designee in relation to their HCV infection during the study.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (9):
- Russia (9):
  - LLC Medical Company Hepatolog /ID# 212384, Samara, Samara Oblast
  - Professor Pasechnikov Gastroenterology and Pankreatology clinic /ID# 217035, Stavropol, Stavropol Kray
  - A. F. Agafonov Republican Clin /ID# 212381, Kazan', Tatarstan, Respublika
  - South Ural State Medical univ /ID# 212020, Chelyabinsk
  - Clinical Inf. Dis Hospital 1 /ID# 217033, Novosibirsk
  - SIH Orlovskiy region city hospital named after S.P. Botkin /ID# 212383, Oryol
  - Perm Regional Center of Cepato /ID# 213992, Perm
  - Saint-Petersburg AIDS Center /ID# 212380, Saint Petersburg
  - Samara State Medical Universit /ID# 217029, Samara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/glecaprevir_pibrentasvir_P19-454.pdf